CLINICAL TRIAL: NCT05743816
Title: Neonatal Antimicrobial Resistance and Outcome (neoAMRO)
Brief Title: Neonatal Antimicrobial Resistance and Outcome
Acronym: neoAMRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: Antibiotic Research UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019.0048
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Neonatal Infection
Keywords: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentre observational study involving NNUs across the UK. Study personnel (Neonatologists and research Nurses) from these NNUs will identify eligible babies in whom a positive culture has been obtained.

This study will help identify the infections leading to death in babies on UK neonatal units, define the clinical characteristics of babies dying from infections, and describe the management of babies dying from infections with a specific focus in their antimicrobial treatment.

DETAILED DESCRIPTION:
The neonIN surveillance network captures data on episodes of invasive neonatal infection on a web-based database. Over 30 UK neonatal units currently contribute to this database in real-time. An episode of neonatal infection is defined as a positive culture collected from a normally sterile site such as the blood, cerebrospinal fluid (CSF) or urine (via catheter or suprapubic aspirate) for which clinicians prescribed at least five days of appropriate antibiotics. Clinical, demographic and microbiological data (including antimicrobial susceptibilities) are collected using a standardised online questionnaire. Denominator data regarding the total number of live-births and neonatal-admissions are collected for each neonatal unit.

Through our study we aim to understand and describe better those infections and risk factors that lead to death. The case-control study will enable us to determine if gaps in optimal management, such as the wrong antibiotic or the wrong dose, are associated with poor outcomes. We can then translate such information into practice and develop / improve clinical guidance in order to improve outcomes.

For the purpose of this study, we will request information on the baby's status (alive/died/not known) at 28 days after the positive culture was obtained. If the baby is alive, then this baby becomes eligible as a control. If the baby has died, then further details will be sought including the date of death and whether death was attributed to the infection.

ELIGIBILITY:
Inclusion criteria:

• Infants on participating NNUs who have an episode of infection with a positive culture.

Ages: 28 Days to 12 Months | Sex: All
Age Groups: Child
Study Population: Neonatal units
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Identifying infections | 5 years
  To identify the infections leading to death in babies on UK neonatal units
Clinical characteristics | 5 years
  To define the clinical characteristics of babies dying from infections
Management of infections | 5 years
  To describe the management of babies dying from infections with a specific focus in their antimicrobial treatment and the antimicrobial resistance profiles of the relevant organisms

SECONDARY OUTCOMES:
Comparing bacterial infections | 5 years
  In a case-control study we will assess the hypothesis that babies who die from bacterial infections on neonatal units do so because they receive inappropriate antibiotic management. To do this we will compare babies who die from bacterial infections with babies who survive bacterial infections on a range of factors including appropriateness, dose and timeliness of antibiotic use.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Galiza, MD, Principal Investigator — St George's, University of London
Locations (1):
- St George's University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data will be made available to all researchers.
Supporting Information: CSR
Time Frame: Clinical Study Report will be made available in the form of a publication within 6 months of study end date.
Access Criteria: Only team members who have access to the database will be able to view study data for their individual site. Sites can also view reports of the general study on the database. The lead site will have capacity to review the full study data for statistical analysis.